CLINICAL TRIAL: NCT05066763
Title: Parkinson's Foundation Surveys
Status: Recruiting | Type: Observational
Sponsor: Parkinson's Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PF-Surveys-01
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with Parkinson's disease
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — non-interventional

SUMMARY:
Parkinson's Foundation Surveys is an initiative seeking to periodically survey people with Parkinson's disease (PD), their care partners and medical professionals to better understand specific aspects of living with PD.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to be contacted by the Parkinson's Foundation for surveys and any future research opportunities
* Anyone who self-reports that they have a diagnosis of Parkinson's disease
* Care partner of a person with Parkinson's disease
* Any health professional that regularly works with people with Parkinson's disease
* 18 years of age or older

Exclusion Criteria:

* People who report that they do not have a diagnosis of Parkinson's disease, are not a care partner to someone with PD or do not work with people with PD in the health setting
* An individual younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's disease, care partners of people with Parkinson's disease, health professional that treats people with Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Total number of survey respondents | 10 years
  Total number of survey participants who consent into the study

CONTACTS AND LOCATIONS:
Locations (1):
- Parkinson's Foundation, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified and coded survey responses may be shared with other researchers.